CLINICAL TRIAL: NCT07399028
Title: A Single-center, Open-label Study to Characterize Human Skin Changes From Biostimulator Treatments Via Non-invasive Imaging
Brief Title: A Study to Characterize Human Skin Changes From Biostimulator Treatments Via Non-invasive Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.050
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Volume Deficiency in the Mid-Face; Skin Laxity; Photo-aged Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Subjects will be treated for correction of fine lines and wrinkles in the cheek area with Sculptra. Subjects will receive 3 treatments with Sculptra, four weeks apart.
  Interventions: Device: Sculptra®

INTERVENTIONS:
Device: Sculptra® — Sculptra injection will be performed to the cheeks using 25 G needle size. Injections will be performed subdermally, i.e., in the subcutaneous and supraperiosteal region. A maximum of 18 mL (2 vials) of Sculptra will be administered per treatment session with a maximum of 9 mL (1 vial) per cheek, evenly distributed within the treatment area.

SUMMARY:
Adult subjects with moderate-to-severe cheek wrinkles will be treated with Sculptra for correction of fine lines and wrinkles in the cheek area.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 45-65 years old
* Females only
* Subject with moderate-to-severe cheek wrinkles on the GCWS
* Subject with intent to undergo correction of cheek wrinkles on both sides of the face
* Subject who in the opinion of the Investigator would need 3 treatments for optimal clinical outcomes
* Subject willing to be photographed at each visit.
* Subjects willing to stop using current facial skincare products for the duration of the study.
* Subject willing to replace the current facial skincare products with the provided facial skincare products, including cleanser, moisturizer and sunscreen, until study completion.
* Ability to read, understand and give consent for participation in the study.
* Agreement to adhere to the procedures and requirements of the study and to report to the site on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

* Subjects with a history of allergy or hypersensitivity to any ingredient of the treatment products.
* Previous tissue-augmenting therapy, contouring, or revitalization treatment in the face, except lips.
* Previous treatment/procedure in the face in the previous 6 months that, in the Investigator's opinion, would interfere with the study injections and/or study assessments or exposed the study subject to undue risk by study participation, or planning to undergo any of these procedures affecting the treatment area at any time during the study.
* Subjects with any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Structural change in midface post-treatment with a biostimulator compared to pre-treatment assessed by standardized VISIA imaging and optical biopsy imaging | 4 weeks, 8 weeks, 12 weeks, 16 weeks, and 20 weeks after baseline
  Images taken with VISIA imaging system and an imaging system using tomography technology at baseline and post-baseline timepoints will be compared to assess structural changes in cheeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No